CLINICAL TRIAL: NCT05674695
Title: Spanish Academy of Dermatology and Venereology Registry of Atopic Dermatitis Therapy
Acronym: BIOBADATOP
Status: Recruiting | Type: Observational
Sponsor: Fundación Academia Española de Dermatología (Other)
Responsible Party: Sponsor
Other Study IDs: FAE-ATO-2018-02
Record Dates: First submitted 2023-01-02; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine; Methotrexate; dupilumab; Adrenal Cortex Hormones; Omalizumab; baricitinib; upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: Ciclosporin — Any systemic drug used for atopic dermatitis in clinical practice
  Other Names: Methotrexate; Dupilumab; Corticosteroids; Omalizumab; Baricitinib; Upadacitinib; Tralokimumab; Topical corticosteroids

SUMMARY:
The Spanish Registry of Systemic therapy in atopic eczema, BIOBADATOP, assesses drug safety and treatment effectiveness as well as treatment impact on quality of life in children and adults with atopic eczema receiving systemic immuno-modulatory therapies in Spanish daily practice.

The main objectives are:

1. To assess short and long-term safety of systemic therapies (including phototherapy) for atopic eczema (pharmacovigilance).
2. To assess short and long-term effectiveness of systemic therapies, providing a basis for shared decision making and guidelines.

Secondary objectives are:

1. To assess short and long-term safety of topical therapies for atopic eczema.
2. To assess effectiveness of different methods of care, including patient training.
3. To describe atopic dermatitis comorbidities.

ELIGIBILITY:
Inclusion Criteria:

1. Paediatric and adult patients with atopic eczema who due to the severity of their disease and/or impact on quality of life are commencing on or switching to a specific systemic immuno-modulatory agent (e.g. CyA, AZA, MTX or new/biologic treatments) for the first time in their life (might have received others, but not this specific one).
2. Diagnosis of atopic eczema in keeping with the UK/Irish diagnostic criteria.
3. Willingness to comply with all study requirements.

Exclusion Criteria:

1. Insufficient understanding of the study by the patient and/or parent/guardian.
2. Patients who are currently participating in a randomised clinical trial.
3. Intention to move to a different geographical area in a short-term (next 3 months).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population intends to be representative of all atopic dermatitis patients treated with systemic drugs in dermatology clinics in Spain.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Rates of adverse events | through study completion, an average of 3 years
  For each drug or drug type
Relative rate of adverse events | through study completion, an average of 3 years
  Compared to a standard drug ( such as cyclosporine). Crude and adjusted

SECONDARY OUTCOMES:
Change in Eczema Area and Severity Index (EASI) | Change between baseline and 6 months
  EASI is used to measure the extent (area) and severity of atopic eczema.The minimum EASI score is 0 and the maximum EASI score is 72. A higher score means more severe or extended disease.
Change in Patient Oriented Eczema Measure (POEM) | Change between baseline and 6 months
  The Patient Oriented Eczema Measure (POEM) is a tool used for monitoring atopic eczema severity. It focuses on the illness as experienced by the patient. It ranges from 0 to 28, with higher scores meaning worse disease.

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar IMIM, Barcelona
  - Hospital Universitario de Gran Canaria Dr Negrín, Las Palmas
  - Hospital Infanta Leonor, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario y Politécnico la Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No